CLINICAL TRIAL: NCT04400708
Title: The Effect of Postoperative Single-injection Adductor Canal Block for Multimodal Pain Control in Patients Receiving Total Knee Arthroplasty Under Spinal Anesthesia
Brief Title: Single-injection Adductor Canal Block for Total Knee Arthroplasty Under Spinal Anesthesia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Jin-Tae Kim, professor, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2004-253-11
Record Dates: First submitted 2020-05-19; First posted 2020-05-22 (Actual); Last update posted 2023-11-24 (Actual); Status verified 2023-11

CONDITIONS: Total Knee Arthroplasty
MeSH Terms: interventions — Control Groups

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control group (Sham Comparator): normal saline injection
  Interventions: Procedure: control group
- test group (Experimental): 0.5% ropivacaine injection
  Interventions: Procedure: adductor canal block

INTERVENTIONS:
Procedure: adductor canal block — After the end of the surgery, at the arrival of PACU, the patient's leg is prepared and draped in a sterile manner. Assisted by the high-frequency linear ultrasound transducer, we target the mid-thigh level and the 22-gauge/8cm needle is introduced in plain through the sartorius muscle. the correct position for the tip of the needle in the adductor canal is checked and a bolus injection of 0.5% ropivacaine 15ml is given.
  Arms: test group
Procedure: control group — After the end of the surgery, at the arrival of PACU, the patient's leg is prepared and draped in a sterile manner. Assisted by the high-frequency linear ultrasound transducer, we target the mid-thigh level and the 22-gauge/8cm needle is introduced in plain through the sartorius muscle. the correct position for the tip of the needle in the adductor canal is checked and a bolus injection of normal saline15ml is given.
  Arms: control group

SUMMARY:
This study evaluates the effect of the single-injection adductor canal block in patients receiving total knee arthroplasty under spinal anesthesia.

DETAILED DESCRIPTION:
This study aims to evaluate the effect of the single-injection adductor canal block in patients receiving total knee arthroplasty under spinal anesthesia. The effect of the single-injection adductor canal and continuous adductor canal block in patients receiving total knee arthroplasty under general anesthesia has been well established. However, due to the residual effect of spinal anesthesia, the effect of the single-injection adductor canal block needs to be determined. The investigators hypothesize that the single-injection adductor canal block will decrease the total sum of 2h, 6h, 12h, and 24h pain score.

ELIGIBILITY:
Inclusion Criteria:

* adult patients receiving total-knee arthroplasty under spinal anesthesia
* ASA class 1-3

Exclusion Criteria:

* infection at the needle injection site
* hard for pain evaluation
* CRPS patient with lower extremity symptom
* chronic opioid user
* those with side effect to local anesthetics
* those getting revision total-knee arthroplasty or with the previous operation at the same knee area
* those getting the surgery under general anesthesia due to the failed spinal anesthesia

Ages: 19 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2020-05-28 (Actual); Primary Completion 2021-06-22 (Actual); Study Completion 2021-06-29 (Actual)

PRIMARY OUTCOMES:
the sum of pain score | 2 hours, 6 hours, 12 hours, and 24 hours after intervention
  VAS pain score (0 to 10) is measured using numeric pain rating scale at 2 hours, 6 hours, 12 hours, and 24 hours 0: no pain, 10: worst pain

SECONDARY OUTCOMES:
Postoperative nausea and vomiting | 2 hours, 6 hours, 12 hours, and 24 hours after intervention
  degree of postoperative nausea and vomiting (0 to 3) 0: no nausea, no vomiting, 1: nausea present, but no vomiting, 2: nausea present, vomiting once, 3: vomiting repeatedly within 30 minutes.
Postoperative opioid consumption | 2 hours, 6 hours, 12 hours, and 24 hours intervention
  amount of postoperative opioid consumption based on oral morphine equivalent daily dose

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Hospital, Seoul, South Korea